CLINICAL TRIAL: NCT02031419
Title: A Phase 1B, Multi-Center, Open-Label Study of Novel Combinations of CC-122, CC-223, CC-292, and Rituximab in Diffuse Large B-Cell Lymphoma and Follicular Lymphoma
Brief Title: Novel Combinations of CC-122, CC-223, CC-292, and Rituximab in Diffuse Large B-cell Lymphoma and Follicular Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Replaced with another clinical trial.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-DLBCL-001
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma, Large B-Cell, Diffuse
Keywords: CC-122; CC-223; CC-292; Rituximab; Lymphoma; Diffuse Large B-Cell Lymphoma; Lenalidomide naïve Follicular Lymphoma; Lenalidomide exposed Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; CC-223; Rituximab; spebrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CC-122 + CC-223 +/- rituximab (Experimental): CC-122 administered orally once daily at 2mg or 3 mg in combination with CC-223 administered orally once daily at 20mg or 30 mg with or without Rituximab administered by IV once every 28 days
  Interventions: Drug: CC-122; Drug: CC-223; Drug: Rituximab
- CC-122 + CC-292 +/- rituximab (Experimental): CC-122 administered orally once daily at 2mg or 3 mg in combination with CC-292 administered orally twice daily at 500 mg with or without Rituximab administered by IV once every 28 days
  Interventions: Drug: CC-122; Drug: CC-292; Drug: Rituximab
- CC-292 + CC-223 +/- rituximab (Experimental): CC-292 administered twice daily at 500 mg in combination with CC-223 administered orally once daily at 20mg or 30 mg with or without Rituximab administered by IV once every 28 days
  Interventions: Drug: CC-223; Drug: CC-292; Drug: Rituximab
- CC-122 + rituximab (Experimental): CC-122 administered orally once daily in combination with Rituximab.
  Interventions: Drug: CC-122; Drug: Rituximab

INTERVENTIONS:
Drug: CC-122 — 2mg or 3 mg administered orally once daily
  Arms: CC-122 + CC-223 +/- rituximab; CC-122 + rituximab
Drug: CC-223 — 20mg or 30mg administered orally once daily.
  Arms: CC-122 + CC-223 +/- rituximab
Drug: Rituximab — 375 mg/m2 administered intravenously once every 28 days
  Arms: CC-122 + CC-223 +/- rituximab; CC-122 + rituximab
Drug: CC-122 — 2mg or 3mg administered orally once daily.
  Arms: CC-122 + CC-292 +/- rituximab
Drug: CC-292 — 500 mg twice a day administered orally.
  Arms: CC-122 + CC-292 +/- rituximab
Drug: Rituximab — 375 mg/m2 administered intravenously once every 28 days
  Arms: CC-122 + CC-292 +/- rituximab
Drug: CC-223 — 20mg or 30mg per day administered orally daily.
  Arms: CC-292 + CC-223 +/- rituximab
Drug: CC-292 — 500 mg twice a day administered orally.
  Arms: CC-292 + CC-223 +/- rituximab
Drug: Rituximab — 375 mg/m2 administered intravenously once every 28 days
  Arms: CC-292 + CC-223 +/- rituximab

SUMMARY:
First study, at multiple clinical centers, exploring the effects of different combinations of compounds (CC-122, CC-223 ,CC-292 and rituximab) to treat Diffuse Large B Cell Lymphoma (DLBCL) and Follicular Lymphoma

DETAILED DESCRIPTION:
Study CC-122-DLBCL-001 is a Phase 1b dose escalation and expansion clinical study of CC 122, CC-223 and CC-292 administered orally as doublets with or without rituximab, in participants with relapsed/refractory DLBCL who have failed standard therapy.

In expansion phase, selected combination will be administered to lenalidomide naïve FL participants and lenalidomide exposed FL participants in addition to relapsed/refractory DLBCL participants.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 18 years or older, with histologically or cytologically-confirmed either:

  1. Chemo-refractory DLBCL (including transformed low grade lymphoma)
  2. Lenalidomide naïve; relapsed or refractory CD20-positive follicular lymphoma (Grade 1, 2, or 3a) following at least one prior standard systemic treatment regimen including systemic chemo-, immune-; or chemo-immunotherapy and at least one prior line of salvage therapy with no prior exposure to lenalidomide, or double-refractory FL participants with no prior exposure to lenalidomide (FL-1 cohort)
  3. Lenalidomide exposed: relapsed or refractory CD20-positive follicular lymphoma (Grade 1, 2, or 3a) previously treated with at least two cycles of lenalidomide-containing regimen (FL-2 cohort), either as a single agent or in combination
* At least one site of measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1.
* Participants must have the following laboratory values:
* Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L or ≥ 1.0 x 109/L (with bone marrow involvement with DLBCL)
* Hemoglobin (Hgb) ≥ 8 g/dL.
* Potassium within normal limits
* Asparate Aminotransferase/Serum Glutamic Oxaloacetic Transaminase (AST/SGOT) and Alanine Aminotransferase/Serum Glutamic-Pyruvic Transaminase (ALT/SGPT) ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5.0 X ULN if liver tumor is present.
* Serum bilirubin ≤ 1.5 x ULN.
* Estimated serum creatinine clearance of ≥ 50 mL/min
* Participants must have the following laboratory values:

Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L without growth factor support for 7 days (14 days if participants received pegfilgrastim).

* Males enrolled into treatment arms receiving CC-122 must: Agree to abstain from donating sperm while taking IP and for at least 95 days following discontinuation of IP

Exclusion Criteria:

* Symptomatic central nervous system involvement.
* Known symptomatic acute or chronic pancreatitis.
* Persistent diarrhea or malabsorption despite medical management.
* Peripheral neuropathy ≥ grade 2
* Impaired cardiac function or clinically significant cardiac diseases
* Participants with diabetes on active treatment (for participants treated on CC-223 containing arms only)
* Prior autologous stem cell transplant (ASCT) ≤ 3 months before first dose.
* Prior allogeneic stem cell transplant with either standard or reduced intensity conditioning.
* Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks prior to starting study drugs, whichever is shorter.
* Participants who have undergone major surgery ≤ 2 weeks prior to starting study drugs.
* Women who are pregnant or breast feeding. Adults of reproductive potential not willing to employ two forms of birth control.
* Participants with known HIV infection, chronic active hepatitis B or C virus (HBV/HCV) infection.
* Participants with treatment-related myelodysplastic syndrome.
* History of concurrent second cancers requiring active, ongoing systemic treatment.
* Prior treatment with a dual mTORC1/mTORC2 inhibitor (CC-223 arms only) or BTK inhibitor (PCI-32765) (CC-292 arms only). [Prior treatment with rapamycin analogues, PI3K or AKT inhibitors, lenalidomide and rituximab are allowed].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2013-12-18 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Safety | From the time of informed consent, throughout dosing period and for 28 days after the last dose of study drug.
  To determine safety profiles and dose-limiting toxicities of study drug combinations using NCI CTCAE v4.

SECONDARY OUTCOMES:
Efficacy | Every 2-3 months until proof of tumor progression
  Tumor response rates using Cheson Revised Response Criteria for Malignant Lymphoma
Pharmacokinetics - CC-223 and CC-292 interaction | Day 1, Day 15
  Area under the plasma concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (8):
  - Stanford Cancer Center, Stanford, California
  - Yale Cancer Center, New Haven, Connecticut
  - Local Institution - 005, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota
  - Local Institution - 001, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Local Institution - 007, Madison, Wisconsin
- Canada (2):
  - Local Institution - 402, Edmonton, Alberta
  - Local Institution - 400, Toronto, Ontario
- France (3):
  - Local Institution - 102, Bordeaux
  - Local Institution - 101, Lyon
  - Local Institution - 100, Villejuif
- Italy (3):
  - Local Institution - 202, Milan
  - Local Institution - 200, Rozzano (MI)
  - Local Institution - 201, Turin

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html